CLINICAL TRIAL: NCT02498613
Title: A Phase 2 Study of Cediranib in Combination With Olaparib in Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-01097; NCI-2015-01097 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1604017576; 9881 (Other: Yale University Cancer Center LAO); 9881 (Other: CTEP); UM1CA186644 (NIH); UM1CA186689 (NIH)
Record Dates: First submitted 2015-07-14; First posted 2015-07-15 (Estimated); Results first posted 2024-07-30 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Advanced Malignant Solid Neoplasm; Metastatic Lung Non-Small Cell Carcinoma; Metastatic Lung Small Cell Carcinoma; Metastatic Pancreatic Adenocarcinoma; Metastatic Triple-Negative Breast Carcinoma; Pancreatic Ductal Adenocarcinoma; Stage III Breast Cancer AJCC v7; Stage III Lung Non-Small Cell Cancer AJCC v7; Stage III Lung Small Cell Carcinoma AJCC v7; Stage III Pancreatic Cancer AJCC v6 and v7; Stage IIIA Breast Cancer AJCC v7; Stage IIIA Lung Non-Small Cell Cancer AJCC v7; Stage IIIA Lung Small Cell Carcinoma AJCC v7; Stage IIIB Breast Cancer AJCC v7; Stage IIIB Lung Non-Small Cell Cancer AJCC v7; Stage IIIB Lung Small Cell Carcinoma AJCC v7; Stage IIIC Breast Cancer AJCC v7; Stage IV Breast Cancer AJCC v6 and v7; Stage IV Lung Non-Small Cell Cancer AJCC v7; Stage IV Lung Small Cell Carcinoma AJCC v7; Stage IV Pancreatic Cancer AJCC v6 and v7; Triple-Negative Breast Carcinoma; Unresectable Lung Small Cell Carcinoma; Unresectable Pancreatic Adenocarcinoma; Unresectable Pancreatic Carcinoma; Unresectable Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — fluoromisonidazole; cediranib; olaparib; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (cediranib maleate, olaparib) (Experimental): Patients receive cediranib maleate PO QD on day 1. Patients undergoing FMISO scan also receive olaparib PO BID beginning the day after the second FMISO scan and the rest of the patients receive olaparib PO BID beginning day 4 of cycle 1. Cycles repeat every 28 days (35 days for cycle 1) in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: 18F-Fluoromisonidazole; Drug: Cediranib Maleate; Other: Laboratory Biomarker Analysis; Drug: Olaparib; Procedure: Positron Emission Tomography

INTERVENTIONS:
Other: 18F-Fluoromisonidazole — Correlative studies
  Other Names: 18F-MISO; 18F-Misonidazole; FLUOROMISONIDAZOLE F-18; FMISO
Drug: Cediranib Maleate — Given PO
  Other Names: AZD2171; AZD2171 Maleate; Recentin
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281
Procedure: Positron Emission Tomography — Correlative studies
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase II trial studies cediranib maleate in combination with olaparib in treating patients with solid tumors that have spread to other parts of the body (advanced/metastatic) or cannot be removed by surgery (unresectable), including breast cancer, non-small cell lung cancer, small cell lung cancer, and pancreatic cancer. Cediranib maleate and olaparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Cediranib maleate may also block the flow of oxygen to the tumor, and may help make the tumor more sensitive to olaparib.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the objective response rate (ORR) of cediranib (cediranib maleate) plus olaparib in combination in patients with advanced or metastatic solid tumors of the following tumor types: non-small cell lung cancer (NSCLC), triple negative breast cancer (TNBC), pancreatic ductal adenocarcinoma (PDAC), and small cell lung cancer (SCLC).

SECONDARY OBJECTIVES:

I. To assess the safety and tolerability of oral administration of cediranib in combination with olaparib in patients with select advanced solid tumors.

II. To estimate progression free survival (PFS) in each tumor cohort.

EXPLORATORY OBJECTIVES:

I. To estimate the prevalence of the mutations of deoxyribonucleic acid (DNA) repair genes in tumors using the BROCA panel and to correlate tumor regression with mutations status. (Integrated) II. To evaluate changes in tumor hypoxia on cediranib treatment compared to baseline by [F-18] fluoromisonidazole (FMISO) positron emission tomography/computed tomography (PET/CT) in patients with NSCLC.

III. To evaluate levels of angiogenesis/inflammatory markers including VEGF at baseline and on treatment.

IV. To evaluate levels of circulating tumor deoxyribonucleic acid (ctDNA) at baseline and on treatment.

OUTLINE:

Patients receive cediranib maleate orally (PO) once daily (QD) on day 1. Patients undergoing FMISO scan also receive olaparib PO twice daily (BID) beginning the day after the second FMISO scan and the rest of the patients receive olaparib PO BID beginning day 4 of cycle 1. Cycles repeat every 28 days (35 days for cycle 1) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks. Patients who discontinue the study treatment for reasons other than disease progression or withdrawal of consent will continue to be followed every 4 weeks until disease progression, start of new therapy, or death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed, metastatic or unresectable malignancy of the following types: (a) non-small cell lung cancer (NSCLC), (b) triple-negative breast cancer (TNBC; defined by estrogen receptor [ER] < 1%, progesterone receptor [PR] < 1% and HER2 1+ or less by immunohistochemistry [IHC]; if HER-2 expression is 2+, a negative fluorescence in situ hybridization [FISH] testing is required) (c) pancreatic adenocarcinoma (PDAC), or (d) small cell lung cancer (SCLC)
* Must have received at least one line of standard systemic treatment for locally advanced or metastatic disease setting of the respective tumor type; for NSCLC, it is either PD-1/PD-L1 inhibitor, or platinum-containing chemotherapy, or an EGFR tyrosine kinase inhibitor or an ALK inhibitor if sensitizing mutation present; TNBC: platinum-containing chemotherapy; PDAC: fluorouracil (5-FU-), gemcitabine-, or taxane-containing chemotherapy either with or without radiation therapy; SCLC: platinum-containing chemotherapy for limited or extensive stage disease
* Patients must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1
* Toxicities of prior therapy (except alopecia) should be resolved to =< grade 1 as per National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0; patients with long-standing stable grade 2 neuropathy or prior grade 2 treatment-related hypothyroidism requiring treatment, provided free T4 within normal range, may be considered eligible after discussion with the study principal investigator (PI)
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2 (Karnofsky >= 50%)
* Life expectancy of >= 4 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin > 9 g/dL
* Total bilirubin =< 1.5 x the institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN
* Creatinine =< 1.5 x ULN OR
* Creatinine clearance >= 45 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal; the creatinine clearance is calculated using Cockcroft-Gault formula
* A urine protein: creatinine ratio of < 1 or < 1 g protein on 24-hour urine collection
* International normalized ration (INR) within 1.25 x ULN institutional limits, except where a lupus anti-coagulant has been confirmed
* Activated partial thromboplastin time (aPTT) within 1.25 x ULN institutional limits, except where a lupus anti-coagulant has been confirmed
* Patients must be able to tolerate oral medications and not have gastrointestinal illnesses that would preclude absorption of cediranib or olaparib
* Adequately controlled thyroid function defined by free T4 within normal range, with no symptoms of thyroid dysfunction
* Adequately controlled blood pressure (BP) < 140 mmHg (systolic) and < 90 mmHg (diastolic) taken in the clinic setting by a medical professional within 2 weeks prior to starting study; patients with hypertension may be managed with up to a maximum of 3 antihypertensive medications; patients who are on 3 antihypertensive medications are highly recommended to be followed by a cardiologist or blood pressure specialist for management of BP while on protocol
* Patients who have the following risk factors are considered to be at increased risk for cardiac toxicities, and must have documented left ventricular ejection fraction (LVEF) by echocardiogram greater than institution's lower limit of normal (or 55% if threshold for normal not otherwise specified by institutional guidelines) obtained within 3 months

  * Prior treatment with anthracyclines
  * Prior treatment with trastuzumab
  * A New York Heart Association (NYHA) classification of II controlled with treatment
  * Prior central thoracic radiation therapy (RT), including RT to the heart
  * History of myocardial infarction within 12 months (patients with history of myocardial infarction within 6 months are excluded from the study)
* The effects of cediranib and olaparib on the developing human fetus are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 4 months after completion of cediranib and olaparib administration
* Ability to understand and the willingness to sign a written informed consent document
* Age >= 18 years. There is no dosing or adverse event data currently available on the use of cediranib or olaparib in patients < 18 years of age, thus excluding them from enrollment

Exclusion Criteria:

* Patients who have had chemotherapy or RT within 3 weeks prior to start of the study agents, or those who have not recovered from adverse events due to agents administered more than 3 weeks earlier
* Patients should not have received any other investigational agents within the past 4 weeks
* Patients with untreated brain metastases, spinal cord compression, or evidence of symptomatic brain metastases or leptomeningeal disease as noted on computed tomography (CT) or magnetic resonance imaging (MRI) scans should be excluded from this clinical trial, since neurologic dysfunction may confound the evaluation of neurologic and other adverse events (AEs); screening brain MRI (or CT if MRI contraindicated) will be required for patients with recurrent NSCLC, TNBC, or SCLC; brain MRI (or CT if MRI contraindicated) is required for PDAC if clinically suspected by patient's symptoms or neurological exam; should patient found to have brain metastasis, treatment of brain metastasis must precede the participation in this study; for patients with known and treated brain metastases is allowed in this study if they fulfill the following criteria:

  * The lesions have improved or remained stable radiographically and clinically for at least 6 weeks after completion of brain irradiation or stereotactic brain radiosurgery and off steroids for at least 6 weeks
* Patients who have received prior inhibitor of VEGF signaling and a poly (ADP-ribose) polymerases (PARP) inhibitor administered in combination; unless administered in combination, patients who received a prior PARP inhibitor or a prior VEGF-signaling inhibitor agent are allowed after discussing with the PI
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cediranib or olaparib
* Participants receiving any medications or substances that are strong inhibitors or inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) are ineligible; dihydropyridine calcium-channel blockers are permitted for management of hypertension
* Current use of natural herbal products or other complementary alternative medications (CAM) or "folk remedies"
* Patients with concomitant or prior invasive malignancies within the past 3 years; subjects with treated limited stage basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the breast or cervix are eligible
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* History of myocardial infarction within 6 months prior to registration
* History of stroke or transient ischemic attack within 6 months prior to registration
* NYHA classification of III or IV
* Current cardiac arrhythmia requiring concurrent use of anti-arrhythmic drugs
* History of hypertensive crisis or hypertensive encephalopathy within 3 years prior to registration
* Clinically significant peripheral vascular disease or abdominal aortic aneurysm (> 5 cm) or aortic dissection; if known history of abdominal aortic aneurysm with >= 4 cm in diameter, all of the following must be met:

  * An ultrasound (US) within the last 6 months prior to registration will be required to document that it is =< 5 cm
  * Patient must be asymptomatic from the aneurysm
  * Blood pressure must be well controlled as defined in this protocol
* A major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to starting cediranib (percutaneous/endobronchial biopsies are allowed)
* History of bowel obstruction within 1 month prior to starting study drugs
* History of hemoptysis or any significant bleeding within the last 1 month prior to enrollment
* Presence of cavitation of central pulmonary lesion
* History of abdominal fistula, intra-abdominal abscess, or gastrointestinal perforation within the 3 months prior to enrollment
* Patients may not have current dependency on intravenous (IV) hydration or total parenteral nutrition (TPN)
* Patients may not have evidence of coagulopathy or bleeding diathesis; therapeutic anticoagulation for prior thromboembolic events is permitted; the clinical indication for therapeutic anticoagulation must be clearly documented prior to enrollment and must be discussed with the P.I.; given the increases risk of serious bleeding from cediranib, patients who are on greater than or equal to 2 anti-thrombotic agents, including but not limited to anti-platelet agents (non-steroidal anti-inflammatory drugs [NSAIDs]/aspirin, clopidogrel), heparin, low molecular weight heparin (LMWH), warfarin, and a direct thrombin inhibitor, will be excluded
* Patients may not have features suggestive of myelodysplastic syndrome (MDS) or acute myelogenous leukemia (AML) on peripheral blood smear or bone marrow biopsy, if clinically indicated
* Pregnant women are excluded from this study because olaparib and cediranib have the potential for teratogenic or abortifacient effects; due to the fact that there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with olaparib and cediranib, breastfeeding should be discontinued if the mother is treated with cediranib and olaparib
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with cediranib or olaparib; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated; HIV-positive patients with undetectable viral loads and CD4 counts > 300, and not on any antiretroviral therapy may be allowed after discussing with the principle investigator
* Any condition that, in the opinion of the treating investigator would interfere with evaluation of the investigational product or interpretation of subject safety or study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2016-08-31 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2026-04-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph W Kim, Principal Investigator — Yale University Cancer Center LAO
Locations (16):
- United States (14):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
- Canada (2):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Groups:
- NSCLC Cohort: Non-Small Cell Lung Cancer (NSCLC) participant cohort.
- TNBC Cohort: Triple-Negative Breast Cancer (TNBC) participant cohort.
- PDAC Cohort: Pancreatic Ductal Adenocarcinoma (PDAC) participant cohort.
- SCLC Cohort: Small Cell Lung Cancer (SCLC) participant cohort.
Period: Overall Study
Arm/Group | NSCLC Cohort | TNBC Cohort | PDAC Cohort | SCLC Cohort
Started (Participants are enrolled.) | 31 | 39 | 24 | 28
Began Treatment | 29 | 38 | 19 | 27
Completed | 26 | 37 | 19 | 27
Not Completed | 5 | 2 | 5 | 1
Not completed — Tx Initiation Criteria Not Met | 2 | 1 | 5 | 1
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Those eligible and placed on study prior to receiving first dose.
Groups:
- Total: Total of all reporting groups
Arm/Group | NSCLC Cohort | TNBC Cohort | PDAC Cohort | SCLC Cohort | Total
Number analyzed (Participants) | 31 | 39 | 24 | 28 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (7.8) | 50.1 (8.2) | 64.2 (10.9) | 63.2 (9.0) | 59.6 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 39 | 10 | 14 | 77
  Male | 17 | 0 | 14 | 14 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 31 | 35 | 23 | 26 | 115
  Unknown or Not Reported | 0 | 3 | 0 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 24 | 23 | 19 | 24 | 90
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 16 | 5 | 4 | 32
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 10 | 0 | 1 | 12
  United States | 30 | 29 | 24 | 27 | 110
Eastern Cooperative Oncology Group (ECOG) [Count of Participants; unit: Participants] — The ECOG scale ranges from 0 to 5. ECOG 0: Fully active; ECOG 1: Restricted in physically strenuous activity but able to carry out light work or sedentary activities; ECOG 2: Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; ECOG 3: Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; ECOG 4: Completely disabled. Cannot perform any self-care. Totally confined to bed or chair; ECOG 5: Dead.
  Participants
    0 | 7 | 9 | 7 | 5 | 28
    1 | 20 | 29 | 15 | 23 | 87
    2 | 4 | 1 | 2 | 0 | 7
    3 | 0 | 0 | 0 | 0 | 0
    4 | 0 | 0 | 0 | 0 | 0
    5 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Measured by Response Evaluation Criteria in Solid Tumors version 1.1. The exact two-sided 95% confidence interval for the objective response rate will be reported.
Time Frame: Up to 4 weeks after completion of study treatment (Up to 43 months)
Population: Those analyzed for clinical activity.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | NSCLC Cohort | TNBC Cohort | SCLC Cohort | PDAC Cohort
Number analyzed (Participants) | 26 | 37 | 27 | 19
proportion of participants | 0.08 [0.01 to 0.15] | 0.16 [0.09 to 0.24] | 0.26 [0.16 to 0.36] | 0 [NA to NA] — There were no responders in this cohort.

2. Secondary Outcome: Incidence of Adverse Events
Description: Graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The outcome was updated upon results entry to reflect the number of graded adverse events per cohort separated by Grade 3 and Grade 4.
Time Frame: Up to 4 weeks after completion of study treatment (Up to 44 months)
Population: All graded adverse events (serious and non serious).
Measure: Number; unit: Adverse Events
Units Other Than Participants: Adverse Events
Arm/Group | NSCLC Cohort | TNBC Cohort | PDAC Cohort | SCLC Cohort
Number analyzed (Participants) | 29 | 38 | 19 | 27
Number analyzed (Adverse Events) | 787 | 830 | 392 | 624
Adverse Events
  Grade 3 | 60 | 71 | 37 | 61
  Grade 4 | 2 | 1 | 2 | 7

3. Secondary Outcome: Progression-free Survival
Description: This outcome was updated at the time of results entry to include the median PFS and the full range of survival time in months for each cohort. The time frame was updated as well. PFS was calculated as the duration of time from start of treatment to time of progression or death, whichever occurs first, assessed up to 4 weeks after completion of study treatment.
Time Frame: Up to 4 weeks after completion of study treatment (Up to 44 months)
Population: Those with evaluable responses.
Measure: Median (Full Range); unit: months
Arm/Group | NSCLC Cohort | TNBC Cohort | PDAC Cohort | SCLC Cohort
Number analyzed (Participants) | 26 | 37 | 19 | 27
months | 3.8 [0.1 to 13.3] | 3.4 [1.4 to 42.7] | 1.8 [1.8 to 7.5] | 4.0 [0.8 to 14.5]

4. Other Pre Specified Outcome: Prevalence of the Mutations of Deoxyribonucleic Acid (DNA) Repair Genes in Each Tumor Cohort
Description: In the first 20 endpoint-evaluable patients with non-small cell lung cancer and 20 endpoint-evaluable patients with triple negative breast cancer, the exploratory analyses will be done using Fisher's exact tests, Mann-Whitney U tests or McNemar's test depending on the type of data observed.
Time Frame: Up to 2 years
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Changes in Tumor Hypoxia by Imaging
Description: Measured by 18F-fluoromisonidazole positron emission tomography/computed tomography scans (non-small cell lung cancer). For the pre- and post-cediranib therapy outcome analysis, paired t- test or Wilcoxon signed-rank test will be applied for the continuous variables.
Time Frame: Baseline to post-cediranib monotherapy
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Changes in Level of Circulating Tumor Deoxyribonucleic Acid (ctDNA) (All Cohorts)
Description: Will be assessed using paired t- test or Wilcoxon signed-rank.
Time Frame: Baseline to post therapy
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Changes in Levels of Angiogenesis/ Inflammatory Markers (Angiome Panel) (All Cohorts)
Description: Will be assessed using paired t- test or Wilcoxon signed-rank.
Time Frame: Baseline to post-therapy
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 44 months
Description: Data are presented for the safety population- those that received at least 1 dose.
Arm/Group | NSCLC Cohort | TNBC Cohort | PDAC Cohort | SCLC Cohort
All-Cause Mortality (participants affected / at risk) | 4/29 | 1/38 | 7/19 | 1/27
Serious Adverse Events (participants affected / at risk) | 13/29 | 19/38 | 12/19 | 10/27
Other Adverse Events (participants affected / at risk) | 29/29 | 38/38 | 19/19 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NSCLC Cohort (N=29) | TNBC Cohort (N=38) | PDAC Cohort (N=19) | SCLC Cohort (N=27)
ABDOMINAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (5) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
ADULT RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ALTERED MENTAL STATUS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BILIARY OBSTRUCTION (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
BILIARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLURRED VISION (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONFUSION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
DEATH NOS (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
DIARRHEA (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
DISEASE PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DRY MUCOUS MEMORIES (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (3)
EDEMA FACE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EDEMA LIMBS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FEVER (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LUNG INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
MALIGNANT DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MILD REACTIVE GASTROPATHY (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
OBSTRUCTION LEFT NEPHROSTOMY (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OPIOID DEPENDENCE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PAIN (General disorders) | 2 (6) | 1 (1) | 0 (0) | 2 (4)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
PELVIC INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
PROGRESSION OF PANCREATIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PROGRESSIVE DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
REVERSIBLE POSTERIOR LEUKOENCEPHALOPATHY SYNDROME (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
SEIZURE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
SKIN INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUDDEN DEATH NOS (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
TAKATSUBO (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
THROMBOEMBOLIC EVENT (Vascular disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
TUMOR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NSCLC Cohort (N=29) | TNBC Cohort (N=38) | PDAC Cohort (N=19) | SCLC Cohort (N=27)
HYPERPHOSPHATEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 (9) | 4 (6) | 7 (11) | 7 (8)
ABNORMAL BALANCE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABSOLUTE MONOCYTE COUNT INCREA (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACID REFLUX (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACTIVATED PARTIAL THROMBOPLAST (Investigations) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 0 (0) | 4 (4) | 1 (2)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCRE (Investigations) | 1 (2) | 5 (12) | 6 (7) | 10 (16)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 3 (3) | 4 (7) | 9 (11) | 4 (4)
ALLERGIC REACTION (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (2)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
AMNESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANEMIA (Blood and lymphatic system disorders) | 4 (7) | 8 (23) | 6 (10) | 7 (14)
ANGULAR CHELITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANION GAP DECREASED (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
ANISOCORIA (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANOREXIA (Metabolism and nutrition disorders) | 14 (26) | 16 (25) | 10 (14) | 12 (22)
ANXIETY (Psychiatric disorders) | 1 (1) | 4 (4) | 2 (2) | 2 (2)
AORTIC VALVE DISEASE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 2 (2) | 2 (2)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ASCENDING AORTA ANEURYSM (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASCITES (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INC (Investigations) | 2 (5) | 9 (12) | 8 (8) | 8 (17)
AST DECREASED (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
ATAXIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 10 (10) | 5 (5) | 7 (8)
BIBASILAR LUNG INFILTRATE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BICYTOPENIA (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BIFASCICULAR BLOCK (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLOATING (Gastrointestinal disorders) | 2 (2) | 3 (6) | 1 (1) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 5 (5) | 2 (3) | 2 (5) | 2 (2)
BLOOD CARBON DIOXIDE ELEVATED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BLOOD IN VOMIT (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLOOD LACTATE DEHYDROGENASE IN (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLOOD SHOT EYES (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BLURRED VISION (Eye disorders) | 3 (3) | 3 (3) | 1 (1) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRONCHIAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRUISING (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
BUN DECREASED (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
BURN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BURNING MOUTH (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BURNING SENSATION IN LLQ SECON (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BURNING SENSATION LLQ (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CARBON DIOXIDE ELEVATED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CARDIAC TROPONIN I INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHILLS (General disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHRONIC MICROANGIOPATHIC CHANG (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CLOGGED TEAR DUCTS (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CLUBBING OF FINGERNAILS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COGNITIVE DISTURBANCE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 1 (1) | 1 (4) | 0 (0) | 1 (1)
CONFUSION (Psychiatric disorders) | 4 (4) | 2 (2) | 2 (2) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 4 (4) | 11 (12) | 5 (5) | 9 (11)
COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COPD EXACERBATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 5 (7) | 2 (2) | 7 (8)
CRAMPS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CREATININE INCREASED (Investigations) | 8 (17) | 7 (19) | 1 (1) | 8 (18)
CYANOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DECREASED AIR ENTRY RIGHT SIDE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DECREASED ALK PHOS (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DECREASED ANION GAP (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DECREASED APPETITE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DECREASED AST (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
DECREASED BREATH SOUNDS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
DECREASED BUN (BLOOD UREA NITR (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DECREASED CHLORIDE (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DECREASED CREATININE (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DECREASED GFR (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DECREASED HEMATOCRIT (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
DECREASED INR (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DECREASED TOTAL PROTEIN (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DECREASED URINE CREATINIE (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 9 (16) | 7 (7) | 5 (5) | 10 (19)
DELIRIUM (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
DENTAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DENTAL CARIES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEPRESSED LEVEL OF CONSCIOUSNE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 3 (3) | 1 (1) | 3 (4)
DIARRHEA (Gastrointestinal disorders) | 17 (38) | 27 (42) | 9 (13) | 19 (31)
DIVERTICULOSIS COLI (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 7 (14) | 6 (9) | 4 (5) | 7 (7)
DIZZINESS (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
DM TYPE II (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DOUBLE VISION (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DRY EYE (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
DRY MOUTH (Gastrointestinal disorders) | 4 (4) | 4 (4) | 3 (3) | 4 (4)
DRY MUCOUS MEMBRANES (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0) | 1 (1) | 4 (4)
DYSESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 8 (12) | 4 (5) | 0 (0) | 4 (4)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1) | 2 (2)
DYSPHONIA (General disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 12 (16) | 3 (3) | 4 (8)
E. COLI BATEREMIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EAR PAIN (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
EARLY SATIETY (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EDEMA FACE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EDEMA LIMBS (General disorders) | 3 (3) | 2 (2) | 3 (7) | 2 (2)
EDEMA TRUNK (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EJECTION FRACTION DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
ELEVATED BUN (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
ELEVATED CARBON DIOXIDE (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
ELEVATED GFR (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ELEVATED HEMATOCRIT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
ELEVATED MCH (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ELEVATED MCHC (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ELEVATED MCV (Investigations) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
ELEVATED MPV (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
ELEVATED NT-PRO BNP (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ELEVATED RDW (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ELEVATED TSH (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
ELEVATED URINE CREATININE (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
ELEVTED HEMATOCRIT (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EOSINOPHIL COUNT INCREASE (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
ERYTHEMA LOWER ABDO GRAFT SCAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
ERYTHEMA LOWER CHEST GRAFT SCAR (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ERYTHEMA/TENDERNESS OVER PORT (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
ERYTHRODERMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ESOPHAGEAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ESOPHAGITIS (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
EYE CRUSTING AND DRAINAGE (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EYE PAIN (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FACIAL MUSCLE WEAKNESS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FACIAL PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 3 (5)
FATIGUE (General disorders) | 18 (32) | 17 (24) | 15 (23) | 13 (22)
FECAL INCONTINENCE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FEELING HOT (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FEVER (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
FEVER BLISTER (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FINGERTIPS NUMBNESS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
FLU LIKE SYMPTOMS (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
FLUSHING (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GAIT DISTURBANCE (General disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
GAS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTEROENTERITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTROENTERITIS (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
GASTROESOPHAGEAL REFLUX DISEAS (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (3) | 3 (3)
GUMS BLEEDING (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GYNECOMASTIA (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HALLUCINATIONS (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 7 (12) | 13 (13) | 4 (4) | 4 (4)
HEARING IMPAIRED (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEART FAILURE (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
HEMATOCRIT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEMATOMA (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEMATURIA (Renal and urinary disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
HEMOGLOBIN INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
HEMOGLOBINURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
HEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HEMOTHORAX (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEPATOMEGALY (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HERPES SIMPLEX RECURRENCE (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HIATAL HERNIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 7 (7) | 2 (4) | 3 (8)
HOT FLASHES (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
HYPERBILIRUBINEMIA (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 1 (2) | 1 (1)
HYPERCOAGUABLE STATE (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 4 (8) | 5 (8) | 8 (9) | 4 (14)
HYPERKALEMIA (Metabolism and nutrition disorders) | 2 (2) | 4 (7) | 4 (5) | 6 (7)
HYPERNATREMIA (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
HYPERPHOSPHATEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (3) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 10 (16) | 26 (38) | 13 (16) | 15 (25)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 11 (15) | 7 (14) | 5 (7) | 6 (10)
HYPOBILIRUBINEMIA (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 3 (4) | 2 (2) | 2 (3) | 2 (3)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOKALEMIA (Metabolism and nutrition disorders) | 4 (8) | 7 (8) | 2 (2) | 4 (6)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 5 (7) | 5 (7) | 1 (1) | 2 (4)
HYPONATREMIA (Metabolism and nutrition disorders) | 7 (11) | 7 (11) | 4 (5) | 10 (14)
HYPOPARATHYROIDISM (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 4 (9) | 5 (6) | 0 (0) | 9 (17)
HYPOTENSION (Vascular disorders) | 1 (2) | 1 (1) | 1 (1) | 2 (2)
HYPOTHYROIDISM (Endocrine disorders) | 3 (4) | 3 (4) | 0 (0) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
INCREASED CARBON DIOXIDE (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INCREASED MCH (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INCREASED MCV (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
INCREASED RDW (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INCREASED RED CELL DISTR (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INR INCREASED (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
INSOMNIA (Psychiatric disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
INTERMITTENT DIARRHEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INTRACRANIAL ATHEROSCLEROSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INTRACRANIAL CAROTID ATHEROSCL (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
JOINT RANGE OF MOTION DECREASE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
KYPHOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LARYNGEAL HEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LEFT ANTERIOR FASCICULAR BLOCK (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LEFT CHEST WALL GRAFT SITE INF (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LEFT CHEST WALL RECONSTRUCTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LEFT EYE CYST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LEFT EYE PTOSIS (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LEFT UPPER CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LETHARGY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
LIP SORE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LIPASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
LIVEDO RETICULARIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LOOSE BOWEL MOVEMENTS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
LOOSE STOOLS (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
LOW ANION GAP (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
LOW AST (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LOW CHLORIDE (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LOW GFR (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LOW MCHC (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LOW RBC (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
LOW TOTAL PROTEIN (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
LOW URINE CREATININE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LUNG INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
LYMPHEDEMA (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 7 (10) | 11 (25) | 6 (11) | 5 (13)
MALAISE (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
MCV INCREASED (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
MCV INCREASED (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
MEAN PLATELET VOLUME INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MEMORY IMPAIRMENT (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MENSES BLEEDING (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MILD STENOSIS AT ORIGIN OF L I (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MITRAL VALVE DISEASE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MOUTH SENSITIVITY (General disorders) | 2 (8) | 2 (6) | 0 (0) | 0 (0)
MOUTH SENSITIVTY (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MOUTH SORE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MOUTH TENDERNESS (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MPV INCREASED (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MPV INCREASED (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
MUCOSITIS ORAL (Gastrointestinal disorders) | 3 (8) | 13 (19) | 0 (0) | 5 (8)
MUSCLE ACHING (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUSCLE CRAMPS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCLE PAIN (NECK) (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (4)
MUSCLE WEAKNESS RIGHT-SIDED (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
MUSCLE WEAKNESS UPPER LIMB (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3) | 1 (1) | 2 (2)
NAIL DISCOLORATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 2 (2) | 0 (0) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 16 (22) | 20 (30) | 7 (10) | 16 (25)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
NEURALGIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1) | 6 (7) | 1 (1) | 1 (1)
NEUTROPHILIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 2 (3) | 2 (2) | 0 (0) | 2 (2)
NUMBNESS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NUMBNESS OT RIGHT NECK AND LEG (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ORAL BURNING WITH HER TOOTHPAS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ORAL PAIN (Gastrointestinal disorders) | 6 (8) | 2 (4) | 1 (1) | 3 (5)
ORAL ULCER (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OROPHARYNGEAL LESIONS (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OROPHERYGEAL LESIONS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ORTHOPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
PAIN (General disorders) | 6 (12) | 7 (10) | 5 (8) | 6 (7)
PAIN DIRECTLY BELOW SHOULD BLADE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 (5) | 8 (11) | 2 (2) | 5 (6)
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PALMAR-PLANTAR ERYTHRODYSESTHE (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (9) | 0 (0) | 3 (6)
PALPITATIONS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
PARESTHESIA (Nervous system disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
PARONYCHIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 4 (4) | 6 (6) | 4 (5)
PHOTOPHOBIA (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PHOTOSENSITIVITY (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
PLANTAR FASCITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 4 (5) | 8 (16) | 8 (13) | 8 (14)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 3 (3) | 1 (1)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PLUGGED EARS (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
PORTAL HYPERTENSION (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
POST OBSTRUCTIVE PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
PREDIABETES (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PRESBYLARYNGIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 2 (4) | 3 (4) | 2 (2) | 2 (2)
PROXIMAL MUSCLE MYOPATHY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PRURITIC RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 2 (2) | 0 (0)
PULMONARY EMBOLISM (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMOBLISM (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PULMONARY VALVE DISEASE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RASH (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (5) | 1 (1) | 5 (5)
RASH PUSTULAR (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RATTLING IN CHEST (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RBC DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RDW INCREASED (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RDW INCREASED (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
REDDENED HANDS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
REDNESS TO RIGHT HAND (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RHINORHEA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RHINORRHEA (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RHINORRHEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RIGHT BUNDLE BRANCH BLOCK (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RIGHT EYE INTERMITTENT BLINDNE (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RIGHT HEART STRAIN (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RIGHT HIP PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RIGHT KNEE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RIGHT RIB PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ROSACEA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RUNNY NOSE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SCAB ON LEFT SIDE OF FACE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SCAB ON RIGHT SIDE OF FACE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SCALING OF PALMS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SCRATCHY THROAT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SEATBELT IRRITATION CAR ACCIDE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SEATBELT IRRITATION FROM ACCID (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SEIZURE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SEPTAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SINUS PAIN (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 3 (4) | 4 (5) | 1 (2) | 1 (1)
SINUSITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
SKIN AND SUBCUTANEOUS TISSUE D (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
SKIN INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SKIN PEELING (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN REDNESS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
SKIN ULCERATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
SMALL FISSURE AT LEFT NARE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SMALL LUMP ON LEFT LOWER CHEEK (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SMALL WOUND RIGHT ANTECUBE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 0 (0) | 4 (4)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUPERIOR VENA CAVA SYNDROME (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
THROAT PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
THROMBOEMBOLIC EVENT (Vascular disorders) | 2 (5) | 3 (3) | 3 (3) | 1 (1)
THROMBOTIC THROMBOCYTOPENIC PU (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
THRUSH (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TINNITUS (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TOTAL PROTEIN DECREASED (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
TRICUSPID VALVE DISEASE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TUMOR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 4 (4) | 3 (3) | 0 (0) | 2 (2)
URETHRAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URINARY FREQUENCY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URINARY HESITANCY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 6 (7) | 0 (0) | 1 (1)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
URINARY TRACT PAIN (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URINE CREATININE DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINE DISCOLORATION (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VAGINAL BLEEDING (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
VAGINAL DRYNESS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VASCULAR ACCESS COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VOCAL CORD PARALYSIS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VOICE ALTERATION (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2) | 0 (0) | 2 (2)
VOMITING (Gastrointestinal disorders) | 16 (21) | 17 (34) | 5 (7) | 7 (13)
WEAKNESS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
WEIGHT LOSS (Investigations) | 13 (19) | 9 (17) | 4 (4) | 9 (18)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
WHITE BLOOD CELL DECREASED (Investigations) | 4 (14) | 11 (26) | 4 (6) | 5 (8)
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
YEAST INFECTION (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT02498613/Prot_SAP_000.pdf